CLINICAL TRIAL: NCT05121558
Title: A Randomized Phase III Clinical Trial of Yoga for Chemotherapy-induced Peripheral Neuropathy Treatment (YCT)
Brief Title: The Effect of Yoga on Nerve Pain Caused by Chemotherapy (Chemotherapy-Induced Peripheral Neuropathy)
Acronym: YCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ting Bao, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-517; R01CA251470 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2021-11-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Nerve Pain; Neuropathy; Neuropathy, Painful; Pain; CIPN - Chemotherapy-Induced Peripheral Neuropathy; Chronic Pain
Keywords: Yoga; Chemotherapy-induced Peripheral Neuropathy; Neuropathic Pain; Pain Management; Dana-Farber Cancer Institute; Memorial Sloan Kettering Cancer Center; Cancer survivor; CIPN
MeSH Terms: conditions — Neuralgia; Neuropathy, Painful; Pain; Chronic Pain; Agnosia | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: 3-arm parallel randomized controlled trial (RCT) comparing yoga to a non-physical education control (EC) and usual care.
Who Masked: Care Provider, Investigator
Masking Description: The PI and investigators will be blinded to the patient's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga (Experimental): Participants will receive twice weekly yoga over the course of 8 weeks.
  Interventions: Other: Yoga
- Education control (EC) (Experimental): Participants will receive twice weekly education over the course of 8 weeks
  Interventions: Other: Education control
- Usual care (UC) (Active Comparator): 8 weeks of usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Yoga — Participants will have instructional yoga classes twice each week over the course of 8 weeks. Each yoga class will be 60 minutes, and it will be taught by an experienced yoga instructor. Participants will be provided with a home-based guided program for days classes are not held. Participants in the yoga group will also have the option to participate in a recorded final check-in session after they have completed their 16 yoga classes. The discussion facilitator will follow the Semi-Structured Interview Guide to further understand participants' experiences in the yoga group.
  Arms: Yoga
Other: Education control — Participants will have educational sessions over 8 weeks. The sessions will be on the causes and impact of Chemotherapy-Induced Peripheral Neuropathy (CIPN), how yoga may help with CIPN, and how different therapies may help with CIPN. To encourage participation and adherence, patients in the EC group will receive sixteen free yoga sessions after completing the study. Patients in the EC group will be asked to not go for their own yoga classes locally until their participation in the study is completed.
  Arms: Education control (EC)
Other: Usual care — Participants in the usual care control group will complete the same assessments as the other two arms. To encourage participation and adherence, patients in the UC group will receive sixteen free yoga sessions after completing the study. Patients in the UC group will be asked to not go for their own yoga classes locally until their participation in the study is completed.
  Arms: Usual care (UC)

SUMMARY:
The purpose of this study is to test whether yoga can reduce nerve pain caused by cancer treatment (chemotherapy-induced peripheral neuropathy, or CIPN). Participants will take one of three approaches:

* Yoga classes
* Educational sessions on the causes and impacts of CIPN, how yoga may help with CIPN, and how different therapies may help with CIPN
* Usual care with standard-of-care medications for CIPN

The researchers will compare how these different approaches affect participants' balance, their risk of falls, and their quality of life. This study will also measure how much yoga can help the reduced sense of touch caused by CIPN.

The functional assessments Timed Up and Go (TUG) and Chair to Stand (CTS) can be safely completed either virtually and in-person and will be mandatory for all patients. The functional assessment Functional Reach Test (FRT) and Quantitative Sensory Testing (QST) assessments that can only be completed in-person are optional at these time points.

ELIGIBILITY:
Inclusion Criteria:

* English-proficient men and women aged ≥18 years
* Free of oncologic disease or or stable disease by clinical examination and history
* Completed neurotoxic chemotherapy such as platinum agents, taxanes, vinca alkaloids, and bortezomib at least three months prior to enrollment
* Diagnosis of CIPN based on symptom history, loss of deep tendon reflexes, or the presence of symmetrical stocking-glove pain, numbness, or paresthesia Grade ≥1 sensory pain based on the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* Self-reported moderate to severe CIPN pain, as defined by a score of 4 or greater on the BPI-SF average pain item over the past week
* On a stable regimen (no change in three months) if taking anti-neuropathy or other pain medications and not taking acetyl-L-carnitine
* Willing to adhere to requirement that no new pain medication be taken throughout the first 12 weeks of the study period
* Willing to adhere to all study-related procedures, including randomization to one of the three arms
* Patient answers "Yes" to at least one factor in the question: "Do you think your balance, gait, posture, alignment, or flexibility has been affected by your experience of CIPN?"

Exclusion Criteria:

* Patients who have received physical therapy or practiced yoga for CIPN in the past 3 months. As patients who have received physical therapy or practiced yoga in this time period may already be experiencing its benefits, we will exclude such patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
measuring Chemotherapy-Induced Peripheral Neuropathy pain severity after Yoga | up to 24 weeks
  as measured by the Brief Pain Inventory-Short Form (BPI-SF) compared to EC and UC arms at week 8 response choices of 0 ("no pain") to 10 ("pain as bad as you can imagine").

CONTACTS AND LOCATIONS:
Overall Officials: Ting Bao, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu